CLINICAL TRIAL: NCT01364129
Title: The Comparative Effectiveness of Telemedicine to Detect Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Steven L. Mansberger, MD, MPH, Legacy Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NPAIHB O5-P-O5; 1-U-48-DP-002673 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2011-04-27; First posted 2011-06-02 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; Diabetic Retinopathy Screening; Ophthalmic Telemedicine; Comparative Effectiveness Research
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Participants in this group have digital images of their retina captured with a non-mydriatic camera and are encouraged to see an eye care provider yearly.
  Interventions: Procedure: Ophthalmic Telemedicine
- Traditional Surveillance (No Intervention): Participants in this group are encouraged to see an eye care provider each year for a diabetic eye exam.

INTERVENTIONS:
Procedure: Ophthalmic Telemedicine — Participants receiving the intervention have digital images of their retina captured with a non-mydriatic camera. The images are then sent to Devers Eye Institute for review and report generation.
  Arms: Telemedicine

SUMMARY:
This project aims to: 1) evaluate the long-term effectiveness of telemedicine to detect diabetic retinopathy when compared to traditional surveillance methods, 2) identify the health belief factors related to adherence with annual diabetic eye exams, and 3) determine the cost-effectiveness of the telemedicine system from the perspective of the community clinic, the third-party payer, and the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* diabetic, at least 18 years old, patient at a participating health clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants that Receive Annual Eye Exam | Baseline; Change from Baseline at 1 Year, 2 Years, 3 Years, 4 Years, and 5 Years (number of follow-up exams depends on number of years enrolled in the study)
  This outcome measure will be used to determine (1) whether the telemedicine system increases the proportion of participants that receive an annual eye exam, and (2) what health belief factors are associated with adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Mansberger, MD, MPH, Principal Investigator — Legacy Health System, Devers Eye Institute; Thomas M Becker, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Hunter Health Clinic, Wichita, Kansas
  - Yellowhawk Tribal Health Center, Pendleton, Oregon

REFERENCES:
- [Derived] Park DW, Mansberger SL. Eye Disease in Patients with Diabetes Screened with Telemedicine. Telemed J E Health. 2017 Feb;23(2):113-118. doi: 10.1089/tmj.2016.0034. Epub 2016 Jun 21. PMID 27328169
- [Derived] Mansberger SL, Sheppler C, Barker G, Gardiner SK, Demirel S, Wooten K, Becker TM. Long-term Comparative Effectiveness of Telemedicine in Providing Diabetic Retinopathy Screening Examinations: A Randomized Clinical Trial. JAMA Ophthalmol. 2015 May;133(5):518-25. doi: 10.1001/jamaophthalmol.2015.1. PMID 25741666